CLINICAL TRIAL: NCT04568538
Title: The Effect of a Shaken Baby Syndrome Prevention Program on Turkish Mothers' Awareness and Knowledge: A Randomized Controlled Study
Brief Title: The Effect of a Shaken Baby Syndrome Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayla Kaya, Research Assistant Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AkdenizUnv
Record Dates: First submitted 2020-09-17; First posted 2020-09-29 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Shaken Baby Syndrome; Mothers
Keywords: awareness; knowledge; mothers; nursing; shaken baby syndrome
MeSH Terms: conditions — Shaken Baby Syndrome

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled study
Who Masked: Participant
Masking Description: The statistician will be blind in evaluating the results. The intervention and control group will be defined as group 1 and group 2 for statistical analysis. Scales will be evaluated by the researcher who cannot be blinded due to the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Randomization with a sealed envelope will be applied to mothers who have 2-4 months old babies who apply to Akdeniz University Hospital Pediatric Outpatient Clinic for health control and who accept the study. A pre-test application will be made in the intervention group. The Researcher will fill in the Personal Information Form and the Shaken baby syndrome assessment survey at this stage.
  The training prepared to prevent shaken baby syndrome, which was prepared immediately after the end of the pre-test application, will be given to the mothers in the intervention group. The training will be given with mothers using one-to-one face-to-face interview method. Necessary equipment will be provided for training. At the end of the training, the questions of the mothers will be answered and a booklet prepared to prevent shaken baby syndrome will be given and tele-consultancy will be provided for 2 months.
  Interventions: Other: Training program
- Control group (No Intervention): No application will be made to the mothers in the control group after the pre-test application. After 2 months, the final test application will be made. After the last test, the mothers in the control group will be given a training and a booklet prepared to prevent shaken baby syndrome.

INTERVENTIONS:
Other: Training program — A training program and booklet content for the education to be given to mothers includes the following topics.
  * What is shaken baby syndrome and what is its cause?
  * What are the harms caused by shaken baby syndrome?
  * How is shaken baby syndrome understood?
  * What problems can shaken baby syndrome cause?
  * What are the measures to be taken? For the training and the content of the booklet, expert opinion was obtained from 10 academic members who are experts in the field of Child Health. An evaluation form was created for pre-test and post-test measurements. Expert opinions were also received for these forms.
  Mothers of 2-4 months old babies who applied to Akdeniz University Hospital Pediatric Outpatient Clinic for check-up were randomized with a sealed envelope and accepted the study. In this way, intervention and control groups can be determined. After the pre-test is done in the intervention group, 2-month training, booklet and tele-consultancy services will be provided.
  Arms: İntervention group

SUMMARY:
Objective: This randomized controlled study aims to examine whether the education program prepared to prevent shaken baby syndrome has an effect on mothers' knowledge and attitudes.

Method: Simple randomization will be used to evaluate the intervention and control groups. The study will be carried out with 90 mothers babies of 2-4 months, who applied to Akdeniz University Hospital Healthy Child Outpatient Clinic (intervention group: 45, control group: 45). After the pre-test, the mothers in the intervention group will be trained and a booklet will be given. Tele-consultancy service will be provided to mothers during the 2-month follow-up period. After 2 months of follow-up, a post-test will be applied to the mothers in the intervention group. The mothers in the control group will not be intervened after the pretest is applied. A post test will be applied 2 months after the pre-test. After the post-test, the mothers in the control group will be trained and a booklet will be given. Ethics committee approval and institutional permission were obtained for the study. Verbal and written consent will be obtained from the mothers during the data collection phase.

DETAILED DESCRIPTION:
Method: The study will be conducted with 90 mothers with 2-4 months old babies who applied to Akdeniz University Hospital Healthy Children Polyclinic (intervention group: 45, control group: 45). Personal Information Form, Shaken baby syndrome assessment survey will be used to collect data. Simple randomization will be used to evaluate the intervention and control groups. In order to identify mothers in intervention groups, sealed-envelope randomization method will used. Mothers and statistician group will be unaware of the evaluation. The researcher will not be blind because of the role he plays in the research.

Following the pretest, the intervention group will be trained to prevent shaken baby syndrome. Expert opinion was obtained from 10 expert faculty members for the content of the training. After the training, the booklet prepared in line with expert opinions will be given to the mother in the intervention group. The booklet will remain with the mother. Tele-consultancy will be given to the mother for 2 months after the pre-test. The control group will also be tested beforehand and will not be intervened afterwards. 2 months after the pre-test, a post-test will be applied to the control group and training will be given to prevent shaken baby syndrome. A training booklet will be given to the mothers in the control group after the final test.

Statistical analysis will be done using SPSS 23.0 and statistical significance will be set at p <0.05.

Support will be received in the analysis phase of the Statistical Information Unit of Akdeniz University.

ELIGIBILITY:
Inclusion criteria:

Having a baby of 2-4 months, Free from physical or mental disability

Exclusion Criteria:

Unhealthy (mother or baby), Any SBS education in the last 2 years

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Shaken baby syndrome knowledge level | 2-4 months
  The increase in the mother's level of knowledge about shaken baby syndrome is the outcome measure.This increase will be measured with "Shaken baby syndrome assessment survey". This form was developed by researchers. After the forms were developed, expert opinions were received from 10 academic members who are experts in the field of child health. It will be evaluated whether there is a statistically significant increase in the post-test data. Statistical analysis will be done using SPSS 23.0 and statistical significance will be set at p <0.05. Support will be received in the analysis phase of the Statistical Information Unit of Akdeniz University.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla KAYA, Dr., Study Director — Akdeniz University, Faculty of Nursing
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rideout L. Nurses' Perceptions of Barriers and Facilitators Affecting the Shaken Baby Syndrome Education Initiative: An Exploratory Study of a Massachusetts Public Policy. J Trauma Nurs. 2016 May-Jun;23(3):125-37. doi: 10.1097/JTN.0000000000000206. PMID 27163220
- [Background] Bechtel K, Le K, Martin KD, Shah N, Leventhal JM, Colson E. Impact of an educational intervention on caregivers' beliefs about infant crying and knowledge of shaken baby syndrome. Acad Pediatr. 2011 Nov-Dec;11(6):481-6. doi: 10.1016/j.acap.2011.08.001. Epub 2011 Sep 21. PMID 21940233
- [Background] Fujiwara T, Yamada F, Okuyama M, Kamimaki I, Shikoro N, Barr RG. Effectiveness of educational materials designed to change knowledge and behavior about crying and shaken baby syndrome: a replication of a randomized controlled trial in Japan. Child Abuse Negl. 2012 Sep;36(9):613-20. doi: 10.1016/j.chiabu.2012.07.003. Epub 2012 Sep 4. PMID 22954642
- [Background] Lynoe N, Elinder G, Hallberg B, Rosen M, Sundgren P, Eriksson A. Insufficient evidence for 'shaken baby syndrome' - a systematic review. Acta Paediatr. 2017 Jul;106(7):1021-1027. doi: 10.1111/apa.13760. Epub 2017 Mar 1. PMID 28130787
- [Background] Squier W. The "Shaken Baby" syndrome: pathology and mechanisms. Acta Neuropathol. 2011 Nov;122(5):519-42. doi: 10.1007/s00401-011-0875-2. Epub 2011 Sep 24. PMID 21947257
- [Background] Narang SK, Estrada C, Greenberg S, Lindberg D. Acceptance of Shaken Baby Syndrome and Abusive Head Trauma as Medical Diagnoses. J Pediatr. 2016 Oct;177:273-278. doi: 10.1016/j.jpeds.2016.06.036. Epub 2016 Jul 22. PMID 27458075
- [Derived] Kaya A, Celik D, Efe E. The effect of a shaken baby syndrome prevention program on Turkish mothers' awareness and knowledge: A randomized controlled study. J Spec Pediatr Nurs. 2022 Apr;27(2):e12369. doi: 10.1111/jspn.12369. Epub 2022 Feb 3. PMID 35118794